CLINICAL TRIAL: NCT00704743
Title: A Prospective Randomized Controlled Trial Comparing Circumferential Casting Versus Splinting in Displaced Colles' Fractures
Brief Title: A Trial Comparing Circumferential Casting Versus Splinting in Displaced Colles' Fractures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Dr. Robert Stenstrom, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P98-0172
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2008-06-25 (Estimated); Status verified 2008-06

CONDITIONS: Colles' Fracture
Keywords: Colles fracture treatment; Displaced fracture of distal radius; distal radius fracture treatment; RCT; Emergency Department; cast; splint; treatment
MeSH Terms: conditions — Colles' Fracture; Emergencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Cylindrical cast
  Interventions: Device: Cylindrical cast
- 2 (Active Comparator): Modified sugar tong cast
  Interventions: Device: Modified sugar tong cast
- 3 (Active Comparator): Volar dorsal splint
  Interventions: Device: Volar dorsal splint

INTERVENTIONS:
Device: Cylindrical cast — Arm cast/immobilization technique for wrist fracture
  Arms: 1
Device: Modified sugar tong cast — Arm cast/immobilization technique for wrist fracture
  Arms: 2
Device: Volar dorsal splint — Arm cast/immobilization technique for wrist fracture
  Arms: 3

SUMMARY:
Displaced fractures of the distal radius requiring closed reduction (otherwise known as Colles fractures) are common in the emergency department. The purpose of the study is to determine if there is any difference between 3 methods of immobilization for these fractures: circumferential cast, volar-dorsal splint, and modified sugar tong splint. Maintenance of position was assessed at 4 weeks after the injury and wrist strength and function were assessed at 2 months and 6 months. We hypothesize that there will not be a clinically important difference between these methods of immobilizing for displaced fractures of the distal radius requiring closed reduction.

Extended description of the protocol, including information not already contained in other fields.

Objectives:

Primary: To determine the effectiveness of three immobilization methods (circumferential cast [CC], volar dorsal splint [VDS], modified sugar-tong [MST] splint) in maintaining the position of displaced distal radius fractures after successful closed reduction.

Secondary to assess long term functional outcomes associated with fiberglass splint immobilization versus standard cylindrical casting in patients maintaining initial non-operative reductions.

Design: Randomized prospective single blind controlled trial Patients/Participants: Patients over 18 years of age who presented to the emergency department with a displaced fracture of the distal radius, requiring closed reduction.

Outcome Measurements: Loss of reduction (radiological slippage or the need for surgical fixation during the 3-4 week primary immobilization period after initial successful reduction). Secondary outcomes were DASH score, return to work, activities of daily living (ADL), wrist pain, range of motion (ROM) and grip strength.

Study Phase Phase 3 Study Type Interventional - Assigned to treatment Recruitment status Completed 2003 Record Verification Date March 2003 Anticipated trial start date November 1998 Last Follow-Up Date December 2002 Data Entry Closure Date January 2004 Study Completion Date July 2004 Purpose Treatment Allocation Randomized

Masking Single Blind Control Active Assignment Parallel Endpoints Efficacy Primary outcome Radiologic slippage of fracture at 4 weeks post reduction

Key secondary outcomes Functional outcomes: DASH score, return to work, activities of daily living (ADL), wrist pain, range of motion (ROM) and grip strength

DETAILED DESCRIPTION:
Primary: To determine the effectiveness of three immobilization methods (circumferential cast [CC], volar dorsal splint [VDS], modified sugar-tong [MST] splint) in maintaining the position of displaced distal radius fractures after successful closed reduction.

Secondary to assess long term functional outcomes associated with fiberglass splint immobilization versus standard cylindrical casting in patients maintaining initial non-operative reductions.

Design: Randomized prospective single blind controlled trial Patients/Participants: Patients over 18 years of age who presented to the emergency department with a displaced fracture of the distal radius, requiring closed reduction.

Outcome Measurements: Loss of reduction (radiological slippage or the need for surgical fixation during the 3-4 week primary immobilization period after initial successful reduction). Secondary outcomes were DASH score, return to work, activities of daily living (ADL), wrist pain, range of motion (ROM) and grip strength.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Displaced fracture of distal radius requiring closed reduction

Exclusion Criteria:

* Open fracture
* Previous displaced fracture involving the same or contralateral distal radius
* neuromuscular deficits or CVA of either upper extremity that impaired functional outcome assessment
* concurrent carpal bone fractures or dislocations - - unstable fractures requiring primary open reduction and internal fixation
* skin allergy or sensitivity to either of the immobilization materials
* Smith's, Barton's or Chauffeur fractures
* Neurovascular compromise of the affected limb - - Bilateral distal radius fractures that prevented follow-up comparison with a normal contralateral limb
* Other significant and concurrent injuries in the ipsilateral extremity.
* Undisplaced distal radius fracture
* Reduction performed in the ED did not meet criteria for successful fracture reduction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 1998-11; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Radiologic slippage of fracture at 4 weeks post reduction | 4 weeks

SECONDARY OUTCOMES:
Functional outcomes: DASH score, return to work, activities of daily living (ADL), wrist pain, range of motion (ROM) and grip strength | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Stenstrom, MD, Ph.D, Principal Investigator — University of British Columbia; Eric Grafstein, MD, Study Director — University of British Columbia
Locations (1):
- Department of Emergency Medicine, St Paul's Hospital, Vancouver, British Columbia, Canada